CLINICAL TRIAL: NCT01447238
Title: Diagnosis of Pancreatic Cysts: Endoscopic Ultrasound With Fine Needle Aspiration (EUS/FNA), Direct Visualization, and Confocal Laser-induced Endomicroscopy-A Pilot Study
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: HS2010-7729
Record Dates: First submitted 2011-07-14; First posted 2011-10-06 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Cysts
Keywords: pancreatic cysts; EUS/FNA; Needle-based Confocal Laser Endomicroscopy (nCLE); fiber optic imaging; EUS/FNA of pancreatic cysts
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Direct visualization and needle based confocal laser-induced endomicroscopy miniprobe — Patients will undergo the EUS-FNA procedure, as per standard of care, plus an additional direct visualization (fiber optic probe) and nCLE procedure with the prototype probes, which will add 10 minutes maximum to the EUS-FNA procedure.
  The probes will be positioned against the lining of the pancreatic cyst, and images will be acquired. After imaging, fine needle aspiration of the lesion will be performed, as usual.
  Other Names: Cellvizio; nCLE; Spyglass

SUMMARY:
The purpose of this study is to assess the yield of combination modalities in the diagnosis of pancreatic cysts using EUS/FNA, Fiber optics (direct visualization probe), and prototype needle based confocal laser-induced endomicroscopy miniprobe (nCLE).

DETAILED DESCRIPTION:
Data will be analyzed descriptively to include patient characteristics, procedural variables, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an EUS-FNA procedure of a pancreatic cyst,
* Aged above 18 years
* Granted written informed consent for the study can be included in the study.

Exclusion Criteria:

* Contraindication for undergoing EUS/FNA procedure (such as unwilling or medically unstable patients, patients with severe coagulopathy, patients with poor visualization on EUS for various reasons, etc)
* Pregnant or breastfeeding
* Allergy to fluorescein
* Renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underoing EUS-FNA procedure for pancreatic cyst.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Assess the yield of combination modalities in the diagnosis of pancreatic cysts using EUS/FNA, Fiber optics (direct visualization probe), and prototype needle based confocal laser-induced endomicroscopy miniprobe (nCLE) | From the date of imaging until follow up for 6 months to two years.
  Data will be analyzed descriptively to include patient characteristics, procedural variables, and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Chang, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Derived] Nakai Y, Iwashita T, Park DH, Samarasena JB, Lee JG, Chang KJ. Diagnosis of pancreatic cysts: EUS-guided, through-the-needle confocal laser-induced endomicroscopy and cystoscopy trial: DETECT study. Gastrointest Endosc. 2015 May;81(5):1204-14. doi: 10.1016/j.gie.2014.10.025. Epub 2015 Jan 26. PMID 25634486